CLINICAL TRIAL: NCT03633019
Title: High-dose Use of Recombinant Human Thrombopoietin in Patients With Moderate or Severe Thrombocytopenia Induced by Chemotherapy
Brief Title: High-dose Use of rhTPO in CIT Patients
Acronym: HUrhTPOCITP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shenyang Pharmaceutical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2018LSK-056
Record Dates: First submitted 2018-08-02; First posted 2018-08-16 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-06

CONDITIONS: Thrombocytopenia
Keywords: thrombocytopenia; rhTPO; real-world study; safety; efficacy
MeSH Terms: conditions — Thrombocytopenia | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- high-dose rhTPO (Experimental): rhTPO (300-600U/kg/day), ih, until the platelets increased by 50 x 109/L compared to the baseline or above 100 x 109/L
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO — high dose rhTPO ih
  Other Names: Recombinant Human Thrombopoietin Injection

SUMMARY:
The research studies the safety and efficacy of high-dose recombinant human TPO in solid tumor patients with moderate or severe thrombocytopenia induced by chemotherapy. Patients with platelet count lower than 50 x 109/L will be enrolled and treated with high-dose rhTPO (300-600U/kg/day) until the platelets increased by 50 x 109/L compared to the baseline or above 100 x 109/L. During the study, the blood routine test will be regularly performed according to the clinical routine (at least once every two days). Finally, the clinical data will be collected and analyzed to validate the efficacy and safety of high-dose rhTPO therapy.

DETAILED DESCRIPTION:
Chemotherapy-induced thrombocytopenia is a common toxic reaction of chemotherapeutic drugs, which may lead to dose reduction, delay or even termination of chemotherapy. Severe thrombocytopenia may cause bleeding and threaten patient's life. rhIL-11 and rhTPO are the only two drugs approved by China Food and Drug Administration for the treatment of chemotherapy-induced thrombocytopenia. The recommended dosage of rhTPO is 300U/kg. Clinical practice in the real world is full of changes and restraints. In the treatment of thrombocytopenia induced by chemotherapy, the actual dose of rhTPO is often below 300U/kg, due to factors such as Specs, economy and convenience. If the dose of rhTPO is insufficient, it can not give full play to the effect and thus can not achieve the purpose of rapid recovery of platelets. Previous clinical studies observed that the effect of rhTPO depends on the given dose. Dosage in the range of 75U-600U/kg of rhTPO were safe in human. While the 75U/kg dose group had no significant effect on the platelet count elevation, the platelet count in other three dose groups of 150U/kg, 300U/kg and 600U/kg increased by 24%, 32%, and 52% (P < 0.01). This research is a real-world study designed to verify the safety and efficacy of high-dose rhTPO in solid tumor patients with moderate or severe thrombocytopenia induced by chemotherapy. Patients with platelet count lower than 50 x 109/L will be enrolled and treated with high-dose rhTPO (300-600U/kg/day) until the platelets increased by 50 x 109/L compared to the baseline or above 100 x 109/L. During the study, the blood routine test will be regularly performed according to the clinical routine (at least once every two days) and the clinical data will be collected and analyzed. It is based on the patient's actual condition and the treatment measure is more consistent with the clinical practice. The results of this study are expected to provide new options and references for clinical treatment of thrombocytopenia induced by chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant solid tumor
* moderate or severe chemotherapy-induced thrombocytopenia, platelet counts less than 50×109/L
* plan to use rhTPO
* be willing to adopt appropriate methods of contraception during the study period and 8 weeks after the end of the study; women of childbearing age must undergo pregnancy tests (serum or urine) within 7 days before entering the study and the result must be negative
* volunteer to participate in the study, sign the informed consent, and cooperate with good compliance

Exclusion Criteria:

* having other diseases that can lead to thrombocytopenia, such as aplastic anemia, myelodysplastic syndrome, leukemia, lymphoproliferative disease, immune thrombocytopenic purpura, thrombotic thrombocytopenic purpura, disseminated intravascular coagulation, thyroid disease, liver cirrhosis, hypersplenism, etc.
* using other non-chemotherapeutic drugs that can cause thrombocytopenia, such as sulfonamides, etc
* with long-term wound or great worry of gastrointestinal bleeding
* with venous thrombosis that need thrombolytic or anticoagulant therapy or high risk of venous thromboembolism
* with infection requiring antibiotic treatment
* History of immunodeficiency, including HIV positive, organ transplantation and other acquired/congenital immunodeficiency disorders
* patients with Hepatitis B(except inactive carrier) or Hepatitis C
* with serious heart disease or cerebrovascular disease
* with heart failure or heart failure history
* with severe anemia that requires long-term use of recombinant human erythropoietin
* congenital thrombocytopenia
* has been used medication for thrombocytopenia
* pregnancy or lactation
* participate in other clinical researchers at the same time
* not suitable to participate in the study in researchers'opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of grade 3 and 4 thrombocytopenia | From time of randomization to the time of platelet counts recover to 75×109/L and above, assessed up to 20days
  Period of time when the platelet counts is lower 75×109/L, days

SECONDARY OUTCOMES:
Adverse event | From randomization until 2 days after treatment completion or withdrawal of patient, whichever comes first, assessed up to 22days
  Any related adverse event during the study according to NCI-CTCAE 4.03, count
Platelets transfusion | From randomization to the time of platelets transfusion, assessed up to 20days
  Platelets transfusion during the study, number of times
platelet count nadir | From randomization to the time of the lowest value of platelets, assessed up to 20days
  the lowest platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiao Zhang, doctor, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China